CLINICAL TRIAL: NCT04120740
Title: Validation of Two Acitivity Monitors in Three Inpatient Populations.
Status: Completed | Type: Observational
Sponsor: Mette Merete Pedersen (Other)
Collaborators: SENS Innovation Aps (Unknown)
Responsible Party: Sponsor-Investigator, Mette Merete Pedersen, Postdoctoral fellow, Copenhagen University Hospital, Hvidovre
Organization: Copenhagen University Hospital, Hvidovre (Other)
Other Study IDs: HH-SENS-FYS-01
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2019-11-21 (Actual); Status verified 2019-11

CONDITIONS: Hip Fractures; Abdominal Surgery; Medical Patients
Keywords: Validility; Activity moitoring
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to investigate the validity of Sens Motion and ActivPAL acitivity monitors. Thirthy-six patients from three different patient populations will be included: 12 acute high-risk abdominal surgery patients (+18 years), 12 hip fracture patients (+65) and 12 older medical patients (+65).

Each patient will be asked to wear two sets of activity monitors while performing a predefined researcher-supervised protocol consisting of a range of positions and activities including lying down, sitting, standing and walking.

Observations measured by time in each position will be used as a golden standard for physical activity and thus compared with the data produced by the acitivity monitors.

DETAILED DESCRIPTION:
The study will investigate the association between activity measured by Sens Motion and ActivPAL acitivity monitors, respectively, and direct observation in order to investigate to which degree the two types of activity monitors are able to classify activity (i.e. lying, sitting, standing, walking, up/down transitions and steps).

Thirty-six patients from three different patient populations will be included: 12 acute high-risk abdominal surgery patients (+18 years), 12 hip fracture patients (+65) and 12 older medical patients (+65). Inclusion criteria to be fullfilled: 1) admission from own home. Patients will be excluded for the following reasons: inability to walk independently with or without a walking aid; inability to transfer from lying to sitting, inability to transfer from sitting to standing, inability to cooperate, and inability to speak or understand Danish.

Each patient will be asked to wear two sets of activity monitors (on the right thigh and on the chest) while performing a predefined, supervised protocol consisting of a range of positions and activities including lying down, sitting, standing and walking.

ELIGIBILITY:
Inclusion Criteria:

* older medical patient (+65)
* older hip fracture patient (+65)
* acute high-risk abdominal surgery patient (+18)
* admitted from own home

Exclusion Criteria:

* inability to walk independently with or without a walking aid
* inability to transfer from lying to sitting and sitting to standing
* inability to cooperate
* inability to understand or speak Danish.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be a convenience sample based on eligible patients from different departments at Copenhagen University Hospital, Hvidovre: Hip fracture patients from the orthopaedic department, patients undergoing acute high-risk abdominal surgery from the department of gastrointestinal surgery, and medical patients from one of four medical departments. The patients will be selected based on the last four digits of their personal identification number.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2019-10-10 (Actual); Primary Completion 2019-11-18 (Actual); Study Completion 2019-11-18 (Actual)

PRIMARY OUTCOMES:
Agreement between classification of activity by activity monitors and direct observation | Approximately 20 minutes
  Agreement between classification of activity by activity monitors and direct observation for lying, sitting, standing, walking, up-down transitions and steps

CONTACTS AND LOCATIONS:
Overall Officials: Mette M Pedersen, Postdoc, Study Chair — Hvidovre University Hospital
Locations (1):
- Copenhagen University Hospital, Hvidovre, Hvidovre, Denmark

REFERENCES:
- [Derived] Pedersen BS, Kristensen MT, Josefsen CO, Lykkegaard KL, Jonsson LR, Pedersen MM. Validation of Two Activity Monitors in Slow and Fast Walking Hospitalized Patients. Rehabil Res Pract. 2022 May 16;2022:9230081. doi: 10.1155/2022/9230081. eCollection 2022. PMID 35615755